CLINICAL TRIAL: NCT00269763
Title: The Clinical Use and Safety of TTS (Fentanyl) in the Management of Pain in Patients With Cancer
Brief Title: Clinical Use and Safety of the Fentanyl Transdermal Therapeutic System (TTS) in the Management of Pain in Patients With Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alza Corporation, DE, USA (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR005983
Record Dates: First submitted 2005-12-22; First posted 2005-12-26 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-04

CONDITIONS: Pain; Cancer
Keywords: patch; pain; fentanyl; narcotic; Cancer
MeSH Terms: conditions — Pain; Neoplasms

INTERVENTIONS:
Drug: Fentanyl Transdermal Therapeutic System (TTS)

SUMMARY:
The purpose of this study is to establish the clinical utility and safety of fentanyl TTS (a transdermal patch delivering the narcotic pain reliever fentanyl) in the treatment of pain in patients with cancer.

DETAILED DESCRIPTION:
This is a single-arm, non-randomized, open-label, multi-center trial to assess the safety and clinical utility of the fentanyl Transdermal Therapeutic System (TTS) for the treatment of pain in patients with cancer. Patients requiring narcotics for pain management are converted from conventional analgesics to oral morphine, and titrated to a stable dose prior to the initiation of fentanyl TTS. The stabilized morphine dose provides the basis for the calculation of the equi-analgesic dose of fentanyl TTS based on established analgesic potency ratios. Patients replace the fentanyl TTS patch every 3 days. Immediate-release morphine is available as rescue medication for breakthrough pain. The adequacy of analgesia, use of morphine rescue medication, and routine safety evaluations are obtained at scheduled intervals throughout the trial.

fentanyl patch

ELIGIBILITY:
Inclusion Criteria:

* Patients currently taking narcotic analgesics for relief of cancer pain
* Able to communicate effectively
* Living with a constant caretaker
* Who have achieved a stabilized morphine dose that provides adequate pain control

Exclusion Criteria:

* Patients with a life expectancy of less than 30 days
* Having history of carbon dioxide (CO2) retention or other cardiac, respiratory or nervous system disease (precludes participation because of the potential for respiratory depression)
* Has severe renal or hepatic insufficiency, active skin disease, a history of allergic reactions to narcotics, or a history of narcotic abuse prior to treatment with narcotics for cancer-related pain
* Has a mental or psychiatric disease
* If female of child-bearing potential, currently pregnant or not practicing an acceptable method contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32
Dates: Start 1987-10; Study Completion 1988-04

PRIMARY OUTCOMES:
Assessment of pain relief; Rescue medication usage

SECONDARY OUTCOMES:
Incidence and severity of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Alza Corporation Clinical Trial, Study Director — Alza Corporation, DE, USA

REFERENCES:
- See also: Clinical use and safety of TTS (fentanyl) in the management of pain in patients with cancer — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=100&filename=CR005983_CSR.pdf